CLINICAL TRIAL: NCT02677571
Title: Thoracic Paravertebral Block Versus Pectoral Nerves Block (Modified PECS) Block in Breast Surgery
Brief Title: PVB vs PECS Block in Breast Surgery
Acronym: PVBvsPECS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituti Ospitalieri di Cremona (Other)
Responsible Party: Principal Investigator, Giorgio Danelli, Chief of the Anaesthesia Department, Istituti Ospitalieri, Cremon, Istituti Ospitalieri di Cremona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20995/2014ps
Record Dates: First submitted 2016-01-23; First posted 2016-02-09 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Reconstruction Breast Surgery
MeSH Terms: interventions — Morphine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PVB (Experimental): 51 patients receiving US guided homolateral paravertebral thoracic block with 30ml of 0.25% levobupivacaine, before general anesthesia (TCI-TIVA).
  Interventions: Procedure: Paravertebral Thoracic block; Drug: Levobupivacaine 0.25%; Drug: Morphine
- PECS (Experimental): 51 patients receiving US guided pectorals nerve block with 30ml of 0.25% levobupivacaine, before general anesthesia (TCI-TIVA).
  Interventions: Procedure: Pectorals nerve block; Drug: Levobupivacaine 0.25%; Drug: Morphine

INTERVENTIONS:
Procedure: Paravertebral Thoracic block
  Arms: PVB
Procedure: Pectorals nerve block
  Arms: PECS
Drug: Levobupivacaine 0.25%
Drug: Morphine

SUMMARY:
Purpose to compare paravertebral thoracic block (PVB) and pectorals nerves block as analgesic option for major breast surgery.

102 patients undergoing reconstruction breast surgery will be randomized into two groups: Group PVB (n=51) will receive US guided paravertebral thoracic block (between T2-T6) performed with 30ml of 0.25% levobupivacaine before general anesthesia (TCI-TIVA) induction.

Morphine patient control analgesia (PCA) with loading dose i.v. titrated by the PACU nurse if pain > 5/10 at rest Group PECS (n=51) will receive US guided pectorals nerves block performed with 30ml of 0.25% levobupivacaine before general anesthesia (TCI-TIVA) induction.

Morphine PCA with loading dose i.v. titrated by the post-anesthesia care unit (PACU) nurse if pain > 5/10 at rest

Primary Outcome Measures:

Morphine consumption (mg) (Time Frame: 24 hours) in two Groups

Secondary Outcome Measures:

Pain at rest and during movement quantified as Numerical Rating Scores (0-10) during the first 24 hours postoperatively.

Eventual side effects such as nausea/vomiting. Time necessary to perform the procedure. Pain during procedure execution quantified as Numerical Rating Scores (0-10) Hypnotic and opioids intraoperative consumption to ensure general anesthesia with Bispectral Index between 40 and 60.

ELIGIBILITY:
Inclusion Criteria:

* age> 18 years
* ASA score I - II - III
* undergoing elective reconstruction breast surgery
* signed informed consent

Exclusion Criteria:

* chronic therapy with opioids/ antidepressants
* urgent/emergent surgery
* postoperative transfer to the intensive care unit
* known allergy to any drug medication
* local skin infection
* epilepsy
* alcohol or drug abuse

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2015-12; Primary Completion 2017-01 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
PCA morphine consumption in the two groups within the first 24 postoperative hours | 24 hours postoperatively

SECONDARY OUTCOMES:
Numerical Rating Scores for pain at rest and during movement | 24 hours postoperatively
Postoperative nausea/vomiting incidence | 24 hours postoperatively
Time of performance | During procedure execution
Propofol consumption in intraoperative period | Intraoperative period
  Propofol consumption in intraoperative period to maintain total intravenous general anesthesia (BIS target 40-60). Propofol consumption in mg/kg/h
Opioids (remifentanyl) consumption in intraoperative period | Intraoperative period
  Opioids (remifentanyl) consumption in intraoperative period to maintain total intravenous general anesthesia (systolic blood pression target: reduction of 20% from base line value). Remifentanyl in mcg/kg/h
Numerical Rating Scores during procedure execution | During procedure execution

CONTACTS AND LOCATIONS:
Overall Officials: Giorgio F Danelli, MD, Study Director — Istituti Ospedalieri di Cremona
Locations (1):
- Azienda Ospedaliera Istituti Ospitalieri di Cremona, Cremona, CR, Italy

IPD SHARING:
Plan to Share IPD: No